CLINICAL TRIAL: NCT04307394
Title: Development of an Adjunctive Video-Based Suicide Prevention Intervention Immediately Following Psychiatric Hospitalization: Open Trial
Brief Title: Development of a Video-based Intervention for Suicide Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1910-001; R34MH119414 (NIH)
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-02

CONDITIONS: Suicide; Psychiatric Hospitalization
Keywords: video intervention; treatment development; open trial
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LifePlans (Experimental): LifePlans is a video series using real patients telling their stories of overcoming suicidal thoughts and behaviors to help others who are struggling with these issues.
  Interventions: Behavioral: LifePlans

INTERVENTIONS:
Behavioral: LifePlans — LifePlans is a video-based intervention, in which patients watch episodes starting during a psychiatric hospitalization and continuing through 1 month post-discharge.

SUMMARY:
The investigators will develop a brief video-based intervention for suicide prevention, called LifePlans. LifePlans will be tested in an initial open trial (n = 10) to examine its feasibility and acceptability. Investigators will recruit patients admitted to a psychiatric hospital for suicidal thoughts and behaviors who will receive the intervention for 4 weeks post-discharge. Patients will be assessed at hospital baseline, 1 month post-discharge, and 6 months post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* current psychiatric hospitalization for suicidal thoughts and behaviors
* 18 years or older
* ability to speak and read English
* plan to continue outpatient treatment
* access to means for viewing videos (computer, tablet, smartphone)

Exclusion Criteria:

* current psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Gaudiano, PhD, Principal Investigator — Butler Hospital; Lisa Uebelacker, Ph.D., Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Upload to NIMH Data Archive
Time Frame: Plan to upload by 7/1/2023

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LifePlans
Started | 10
Completed | 5
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | LifePlans
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.00 (15.67)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 6
  Gender: Male | 1
  Gender: Trans-female | 1
  Gender: Trans-male | 1
  Gender: More than one gender | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: The Client Satisfaction Questionnaire is a self-report measure of patient satisfaction with treatment. The total score will be used and ranges from 8 to 32 with increased scores indicating greater satisfaction with treatment.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LifePlans
Number analyzed (Participants) | 5
score on a scale | 25.00 (5.83)

2. Secondary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia Suicide Severity Rating Scale is an interviewer-rated measure of suicidal thoughts and behaviors. The total score (sum of items) will be used and ranges from 2 to 25 with higher scores indicating higher suicidal thoughts and behaviors.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LifePlans
Number analyzed (Participants) | 5
score on a scale
  Baseline | 13.80 (2.39)
  Month 1 | 13.60 (7.67)
Statistical Analysis 1: Comparison: LifePlans; Test type: Superiority; p = 0.957, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | LifePlans
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LifePlans (N=10)
Re-hospitalization (Psychiatric disorders) | 4 (5)

LIMITATIONS AND CAVEATS:
This is a treatment development study and therefore was not designed to test the efficacy of the intervention given the small sample size. Instead, the goal was to examine feasibility and acceptability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT04307394/Prot_SAP_000.pdf